CLINICAL TRIAL: NCT06953388
Title: SPARK-VNS: Facilitating Adaptive Posttraumatic Processing With Non-Invasive Vagus Nerve Stimulation
Brief Title: Understanding Non-invasive Vagus Nerve Stimulation Effects in PTSD
Acronym: SPARK-VNS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Danielle Taylor, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-23-05-5811
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; brain stimulation; fear learning; autonomics; fear potentiated startle
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS (Experimental): Active transcutaneous auricular vagus nerve stimulation
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham taVNS (Sham Comparator): Active transcutaneous auricular vagus nerve stimulation
  Interventions: Device: sham transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — FDA-cleared Digitimer DS7A Constant Current Stimulator (Digitimer Ltd., USA) will deliver electrical stimulation for 60 mins. Active stimulation will consist of direct electrical stimulation to the inner side of the left tragus (anode on the cymba concha, cathode on the surface of the tragus), thereby stimulating the ABVN. Stimulation parameters will consist of 500μs pulse width, 25Hz frequency, delivered at 200% of each participant's individual perceptual threshold (PT) in 60sec on/off trains.
  Arms: Active taVNS
Device: sham transcutaneous auricular vagus nerve stimulation — FDA-cleared Digitimer DS7A Constant Current Stimulator (Digitimer Ltd., USA) will deliver electrical stimulation for 60 mins. Sham will be delivered to the ear lobe. Stimulation parameters will consist of 500μs pulse width, 25Hz frequency, delivered at 200% of each participant's individual perceptual threshold (PT) in 60sec on/off trains.
  Arms: Sham taVNS

SUMMARY:
The goal of this study is to determine how non-invasive brain stimulation (delivered through the ear called vagus nerve stimulation) affects fear learning processes in people who have experienced psychological trauma. To answer these questions, we measure bodily responses (heart rate, sweat, startle) and questionnaires. The main questions it aims to answer are:

Does non-invasive vagus nerve stimulation help reduce anxious arousal? Does non-invasive vagus nerve stimulation help dampen learned fear?

DETAILED DESCRIPTION:
This study aims to determine how non-invasive brain stimulation (delivered through the ear) affects learning processes. During this study, participants who have experienced a trauma will be asked to complete surveys and come to the lab for about 7 hours across four lab visits. Researchers will measure body responses (heart rate, skin conductance, startle), while the ear is stimulated. Participants also will be asked to complete a startle task. The study is at the Wayne State University Tolan Park Research Clinic. Participants will be compensated for their time. To be eligible, participants must be 18-70 years old, have experienced or witnessed a traumatic event, be able to commit 7 hours of time to the study, and be able to wear sensors on their hands, arms, and head and sit quietly at a computer.

Aim 1. Establish feasibility and acceptability of taVNS in a diverse sample of Detroit metro residents with symptoms of posttraumatic stress. It is hypothesized that taVNS delivery will be feasible and acceptable for individuals with trauma exposure and PTS symptoms, and that there will be no difference in acceptability/tolerability between the active and sham conditions.

Aim 2. Establish the effects of active versus sham taVNS on physiological indicators during fear extinction. It is hypothesized that active compared to sham taVNS will a) result in facilitation of fear extinction, and b) show greater modulation of physiological responding. Exploratory Aim: Data will be explored for individual differences (affective blunting, hyperarousal, impaired discrimination of conditioned stimuli) which moderate taVNS effects.

This proposed project will determine how taVNS delivered at higher doses than have been previously administered influence the course of adaptive posttraumatic processing in a sample with trauma exposure, while evaluating the psychophysiological profile in multiple contexts.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80
2. Fluent in English
3. Experience with a DSM-5 Criterion A trauma (LEC-5)
4. Probable PTSD (PCL-5 ≥ 32)

Exclusion Criteria:

1. Visual or Auditory impairment
2. Major injury at time of screen or study procedures
3. Taking ≥20 mg morphine per day
4. Current substance use or intoxication (12-panel drug test)
5. Intellectual disability (MoCA)
6. Self-inflicted injury
7. Occupational injury
8. Prisoner
9. Ongoing domestic violence
10. Pregnant or breastfeeding
11. Contraindications for taVNS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Fear potentiated startle (FPS) | From enrollment to the end of the cross over visit at week 2
  FPS modulation, an objective behavioral indicator of defensive reactivity, is measured during acquisition and extinction, collected using electromyogram (EMG) of the right orbicularis oculi muscle with the EMG module of the Biopac MP160 for Windows.
Skin Conductance (SC) | From enrollment to the end of the cross over visit at week 2
  SC is measured using the electrodermal activity (EDA) module of the Biopac system. Two disposable pre-gelled Ag/AgCl electrodes are placed on the hypothenar surface of the non-dominant hand. SCR is defined as the increase from SC during a 1s pre-CS+ onset baseline to SC during the 3-6s post-CS+ onset.
Heart Rate (HR) | From enrollment to the end of the cross over visit at week 2
  HR is acquired via electrocardiogram (ECG) Biopac module. Three disposable pre-gelled Ag/AgCl electrodes are used: one each on the right and left sides of the torso, 1cm below the clavicle, and a third on the inside of the left wrist. The HR response is defined as the increase in HR from a 1m baseline prior to the first airblast to 1m after first airblast.
Subjective Units of Distress (SUDS) | From enrollment to the end of the cross over visit at week 2
  SUDS is recorded pre- and post- fear acquisition and extinction, and at baseline and recovery. Arousal measures will be evaluated individually and in combination to determine multivariate effects. SUDS and objective responses will be monitored, as investigations show discordance within and between objective and subjective measures of distress.
  SUDS are on a scale of 0 (no anxiety/distress, calm and relaxed) to 100 (extreme anxiety/distress, worst ever experienced).
Unconditioned Stimulus Expectancy Ratings | From enrollment to the end of the cross over visit at week 2
  Identification of threat/conditioned stimulus with reinforcement (CS+) and safety/conditioned stimulus without reinforcement (CS-) is used to assess US expectancy during fear acquisition and extinction, consistent with mentors', Jovanovic and Norrholm's, research. Individuals respond on a keypad (Cedrus, Inc.) after each trial regarding CS-US contingencies.
  Responses consist of 3 button presses (Yes, No, I don't know) for whether participants believe a shape (CS+/CS-) will be followed by the US.

CONTACTS AND LOCATIONS:
Locations (1):
- Tolan Park Research Clinic, Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
A. Types and amount of scientific data expected to be generated in the project:
  Demographic, end user feedback, clinical (self-report surveys), and physiological data will be collected from 60 individuals with PTSD. Data will be collected, processed, and then shared at the individual level. All data will be de-identified prior to uploading to the repository. However, sufficient information necessary for generating a global unique identifier (GUID) for the NIMH data archive (NDA) will be collected for each subject.
  B. Scientific data that will be preserved and shared, and the rationale for doing so: Scored assessments and self-report surveys will be shared to the NDA, as well as scored physiology measures. Individual, item-level scores, may result in identification of participants, and will not be shared. Any potentially identifiable PHI will be removed from data sets.
  C.Study protocols, data collection instruments, data processing and scoring protocols, and syntax for data analysis.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: A. All data will be deposited to the NIMH data archive (NDA) 12 months after the study begins and will be deposited biannually following the first submission.
  B. Within the first 6 months of an NDA Data Submission agreement will be submitted by the PI through the NDA website, which will allow for access to the NDA Collection page where data will be submitted. The NCT# will be submitted within this agreement. Data will be findable for the research community using the NDA Collection page. An NDA study will be created for each publication and each study will be assigned a digital object identifier (DOI). The DOI will be referenced in the publication so that the research community can access the data used in the publication. C. The research community will have access 1-2 years after study end date. Publication will be linked to a study containing the data used in that publication and may be found using the DOI when the pre-print is available. NDA will determine data preservation duration.
Access Criteria: NDA will control data access. Researchers will submit a data access request for broad use and must be sponsored by an NIH recognized institution and have a research-related need to access the data. The NDA data access committee will make final determination on which requests to grant.
URL: https://nda.nih.gov/